CLINICAL TRIAL: NCT02787135
Title: Efficacy and Mechanisms of Change of an Emotion-oriented Version of Cognitive-behavioral Therapy for Psychosis (CBTp-E) in Reducing Delusions. A Randomized-controlled Treatment Study (CBTd-E)
Brief Title: Efficacy and Mechanisms of Change of an Emotion-oriented Version of Cognitive-behavioral Therapy for Psychosis
Acronym: CBTd-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: University of Hamburg-Eppendorf (Other); Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stephanie Mehl, Prof. Dr. rer. nat., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBTd-E_MehlLincoln2016
Record Dates: First submitted 2016-02-26; First posted 2016-06-01 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia; Psychotic Disorders; Delusions; Emotions; Self-esteem; Sleep
Keywords: Delusions; Schizophrenia; Cognitive Behavior Therapy; Emotion; Emotion regulation; self-esteem; sleep quality; Efficacy of change
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Delusions; Emotional Regulation; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBTd-E (Active Comparator): Experimental: emotion-oriented Cognitive Behavior Therapy focused on delusions for patients with schizophrenia-spectrum disorders and delusions. The therapeutical intervention follows a treatment-manual consisting of two modules. Patients work on two modules every week for 25 weeks in a row. Module I comprises psychoeducation on emotions, training radical acceptance of emotions and mindfulness, cognitive and behavioral strategies in order to change negative emotions and in order to foster positive emotions and suggestions for life-style changes (positive activities, sports, stress reduction). In the second module, the focus is on self-acceptance. Patients receive psychoeducation on self-acceptance and learn strategies in order to reduce negative self-schema and foster positive self-schema.
  Interventions: Behavioral: emotion-oriented Cognitive Behavior Therapy
- Treatment as Usual (Placebo Comparator): Patients who are randomized and assigned to the Wait-list receive treatment as usual (regular visits to a physicist every third month and antipsychotic medication). After six month the waiting list patients receive the treatment specified above.
  Interventions: Behavioral: emotion-oriented Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: emotion-oriented Cognitive Behavior Therapy — Emotion-oriented Cognitive Behavior Therapy with a focus on delusions: Aim of the intervention is to change factors that are involved in the formation and maintenance of delusions: emotional stability and regulation of negative emotions, sleep quality and self-esteem.
  Other Names: CBTd-E

SUMMARY:
The aim of the present single-blind randomized-controlled therapy study is to assess the efficacy of a new form of Cognitive Behavioral Therapy for delusions with a focus on emotion regulation, improvement of self-esteem and sleep quality (CBTd-E).

DETAILED DESCRIPTION:
Numerous meta-analyses have found Cognitive Behaviour Therapy for psychosis (CBTp) to be effective. The effect sizes that are achieved for positive symptoms in addition to antipsychotic treatment vary between small to medium. However, the effect sizes for changes in delusions are somewhat lower. Thus, it could prove beneficial to tailor CBTp interventions more precisely to the processes that are relevant to delusions. Empirically derived models of the formation and maintenance of delusions postulate an important role of cognitive biases, emotional factors and self-esteem. Additional studies have demonstrated the relevance of impaired sleep to delusions. Nevertheless, CBTp interventions that aim to change delusions tend to focus mainly on reasoning bias.

The results of several uncontrolled pilot studies that focused primarily at improving emotional factors, quality of sleep and self-esteem in patients with delusions indicate that changes in these factors have the potential to reduce delusions. However, in these studies the singular interventions were short and were not implemented into a broader therapy rational. It can thus be assumed that a combination of CBT-interventions within a broader therapy rational might have an even greater impact on delusions.

The aim of the present single-blind randomized-controlled therapy study is to assess the efficacy of a new form of Cognitive Behavioral Therapy for delusions with a focus on emotion regulation, improvement of self-esteem and sleep quality (CBTd-E) that will be applied in 25 individual sessions. Moreover, the study aims to test whether the efficacy of CBTd-E is mediated by the postulated processes. The main hypotheses are:

1. Baseline differences: in comparison to healthy controls, patients with schizophrenia show more pronounced problems in emotion regulation, a reduced sleep quality and a lower and less stable self-esteem.
2. Efficacy of CBTd-E: patients with acute delusions who receive CBTd-E show a more pronounced reduction of delusions (primary outcome), as well as a more pronounced reduction of positive symptoms, depression and general psychopathology, a stronger improvement in general and social functioning and will receive lower doses of antipsychotic medication (secondary outcomes) at post-treatment.
3. Mediation: the effect of CBTd-E on change in delusions is mediated by a) improved emotional stability and ability to regulate one's own emotions, b) improved sleep quality, c) improved and more stable self-esteem.

In addition to questionnaires and interviews, behavioral paradigms, psychophysiological assessments and electronic diaries will be used to test the hypotheses. If we can demonstrate that CBTd-E reduces delusions, this would provide us with a more acceptable and feasible therapy for treating delusions.

ELIGIBILITY:
Treatment Group:

Inclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, delusional disorder (DSM-5 diagnosis)
* Delusions present in the last three months (score of at least three in three out of six PSYRATS scores)
* problems in at least two out of three possible mediators: sleep problems (ISI sum score > 7), low self-esteem (score > 3in the BCSS negative self scale) and/or problems in emotion regulation (score in all items < 4)
* fluent in German language
* agree to participate
* estimated general intelligence of at least 70 in the German Mehrfachwahlwortschatztest (MWT-B)
* no present suicidality

Exclusion Criteria:

* acute suicidal tendency
* comorbid diagnosis of borderline personality disorder and/or substance use disorder in the last six month
* taking of Benzodiazepines

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Psychotic Rating Scale (PSYRATS) delusions scale | Change between pre-therapy and post-therapy assessment after six month
  Assessment of delusion frequency, delusion distress, conviction and loss of quality of life due to the delusion

SECONDARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) | Change between pre-therapy and post-therapy assessment after six month
  Assessment of positive, negative and general symptoms of schizophrenia
Change in Calgary Depression Rating Scale for Schizophrenia (CDSS( | Change between pre-therapy and post-therapy assessment after six month
  Assessment of depressive symptoms in patients with schizophrenia
Change in Role Functioning Scale (RFS) | Change between pre-therapy and post-therapy assessment after six month
  Assessment of social functioning
Change in Peters et al. Delusions Inventory (PDI- R) | Change between pre-therapy and post-therapy assessment after six month
  Assessment of self-rated delusion frequency, conviction and distress.

OTHER OUTCOMES:
Change in Emotion-regulation Questionnaire (ERQ) | Change between pre-therapy and post-therapy assessment after six month
  Questionnaire assesses the regular use of emotion regulation strategies
Change in Emotion regulation inventory | Change between pre-therapy and post-therapy assessment after six month
  Questionnaire assesses the regular use of emotion regulation strategies
Change in Paranoia assessed with Electronical mobile assessment | Change between pre-therapy and post-therapy assessment after six month
  Assessment of present emotions, emotion regulation strategies, present symptoms of psychosis, present delusions, self-esteem for six consecutive days (10 assessments per day) in daily life
Change in Sleep quality as assessed with an Actiwatch | Change between pre-therapy and post-therapy assessment after six month
  Assessment of sleep-quality using an electronic bracelet for six consecutive days, sleep quality is assessed with movement detectors and light sensors
Change in Emotion regulation quality as assessed experimental using International Affect Picture System Paradigm for the Assessment of emotion regulation (IAPS) | Change between pre-therapy and post-therapy assessment after six month
  Assessment of effectiveness of use of emotion regulation strategies after experimental induction of fear, assessment of heart rate and skin conduction
Change in heart rate variability | Change between pre-therapy and post-therapy assessment after six month
  Assessment of heart rate variability with sensors during stress induction (reaction experiment) and during rest
Change in Brief Core Schema Scale (BCSS) | Change between pre-therapy and post-therapy assessment after six month
  Assessment of positive and negative self-schemata and schemata on others
Change in Insomnia Severity Index (ISI) | Change between pre-therapy and post-therapy assessment after six month
  The ISI assesses present sleep problems
Change in Self-Compassion Scale (SCS) | Change between pre-therapy and post-therapy assessment after six month
  SCS assesses self-compassion and self-esteem
Change in Self-perception of emotional competencies (SEK-27) | Change between pre-therapy and post-therapy assessment after six month
  Questionnaire assesses the regular use of emotion regulation strategies

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Mehl, Ph. D., Study Chair — Philipps University Marburg; Tania M Lincoln, Ph. D., Study Chair — University of Hamburg-Eppendorf; Tobias Teismann, Ph. D., Principal Investigator — Ruhr University of Bochum
Locations (2):
- Germany (2):
  - University of Marburg, Faculty of Clinical Psychology and Psychotherapy, Marburg, Hesse
  - University of Hamburg, Faculty of Clinical Psychology and Psychotherapy, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kammerer MK, Mehl S, Ludwig L, Lincoln TM. Sleep and circadian rhythm disruption predict persecutory symptom severity in day-to-day life: A combined actigraphy and experience sampling study. J Abnorm Psychol. 2021 Jan;130(1):78-88. doi: 10.1037/abn0000645. Epub 2020 Nov 19. PMID 33211503
- [Derived] Ludwig L, Mehl S, Krkovic K, Lincoln TM. Effectiveness of emotion regulation in daily life in individuals with psychosis and nonclinical controls-An experience-sampling study. J Abnorm Psychol. 2020 May;129(4):408-421. doi: 10.1037/abn0000505. Epub 2020 Feb 27. PMID 32105124